CLINICAL TRIAL: NCT01199094
Title: Clinical Assessment of Patients With High Bone Mass Due to Mutation in Low Density Lipoprotein l Receptor 5
Brief Title: Clinical Assessment of Patients With High Bone Mass Due to Mutation in Lrp5
Status: Completed | Type: Observational
Sponsor: Odense University Hospital (Other)
Responsible Party: Kim Brixen, Professor, consultant, Odense University Hospital
Other Study IDs: LRP5-HBM
Record Dates: First submitted 2010-09-09; First posted 2010-09-10 (Estimated); Last update posted 2010-09-10 (Estimated); Status verified 2010-08

CONDITIONS: Osteopetrosis
Keywords: low density lipoprotein receptor 5; high bone mass; autosomal dominant osteopetrosis type I; bone turnover markers
MeSH Terms: conditions — Osteopetrosis; Osteopetrosis autosomal dominant type 1

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Cross-Sectional
Biospecimen Retention: Samples With DNA — Serum, plasma, DNA as well as fat and skin biopsies
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Patients with mutation in the Lrp5 gene: Patients known to have a mutation in Lrp5 known to be causing a high bone mass phenotype

SUMMARY:
The aim of the study is to describe patients with a high bone mass phenotype due to a mutation in the low density lipoprotein l receptor 5 gene (LRP5) and compare them with age and sex matched controls. Moreover, bone density and microarchitecture as well as markers of bone metabolism are evaluated

DETAILED DESCRIPTION:
Cases and controls are closely matched on age and sex and evaluated cross-sectionally.

Dual x-ray absorptiometry (DXA) and high resolution peripheral quantitative computed tomography (HR-pQCT) are used in order to evaluate bone density as well as microarchitecture. Bone turnover markers and body composition are also measured.

ELIGIBILITY:
Inclusion Criteria:

* Lrp5 mutation/ADOI

Exclusion Criteria:

* Pregnancy

Min Age: 8 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult, Older Adult
Study Population: Case-control study on almost 40 individuals
Sampling Method: Non-Probability Sample
Enrollment: 38 (Actual)
Dates: Start 2009-01; Primary Completion 2010-04 (Actual); Study Completion 2010-06 (Actual)

PRIMARY OUTCOMES:
Bone microarchitecture as assessed by high resolution quantitative computed tomography (HR-pQCT) | 12 weeks
  HR-pQCT is used to evaluate bone microarchitecture, i.e. bone trabeculae, cortical thickness and trabecular number. Aim is to test if the microarchitecture of these patients are different that observed in normal controls

SECONDARY OUTCOMES:
Changes in bone turnover markers | 12 weeks
  Markers of bone resorption and formation are investigated.
Bone mineral density | 12 weeks
  DXA is used to evaluate bone mineral density at total hip, spine, whole body and forearm.

CONTACTS AND LOCATIONS:
Overall Officials: Kim Brixen, Professor, Principal Investigator — Odense University Hospital
Locations (1):
- Odense University Hospital, Osteoporosis Clinic, Odense, Denmark

REFERENCES:
- [Result] Frost M, Andersen TE, Yadav V, Brixen K, Karsenty G, Kassem M. Patients with high-bone-mass phenotype owing to Lrp5-T253I mutation have low plasma levels of serotonin. J Bone Miner Res. 2010 Mar;25(3):673-5. doi: 10.1002/jbmr.44. PMID 20200960